CLINICAL TRIAL: NCT05999812
Title: Phase II Single-arm, Single-center Clinical Trial of All-trans-retinoic Acid, Bevacizumab and Atezolizumab in Refractory Microsatellite Stable Colorectal Cancer
Brief Title: Clinical Trial of All-trans-retinoic Acid, Bevacizumab and Atezolizumab in Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Syed Kazmi, Assistant Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0409
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tretinoin; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): * ATRA orally 45 mg/m2 daily in 2 divided doses days 1-7, repeat every 14 days
  * Atezolizumab IV D1, 840 mg every 14 days
  * Bevacizumab IV D1, 10 mg/kg every 14 days
  Interventions: Drug: all trans Retinoic Acid; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: all trans Retinoic Acid — ATRA orally 45 mg/m2 QD in 2 divided doses days 1-7, repeat every 14 days
  Other Names: Tretinoin; ATRA
Drug: Atezolizumab — Atezolizumab IV D1, 840 mg every 14 days
Drug: Bevacizumab — Bevacizumab IV D1, 10 mg/kg every 14 days

SUMMARY:
The main purpose of this clinical trial is to learn about the good and the bad effects of all trans retinoic acid (ATRA), atezolizumab and bevacizumab as a possible treatment for advanced colorectal patients.

Participants will be treated with the following combination of these drugs:

1. ATRA will be given in a pill form to be taken twice a day at home for 7 days starting on day 1 of a cycle.
2. Atezolizumab will be given through a vein in arm or through mediport over 60-90 minutes every 2 weeks in the outpatient chemotherapy infusion centers at UTSW.
3. Bevacizumab will be given through a vein in arm or through mediport over 20-40 minutes every 2 weeks in the outpatient chemotherapy infusion centers at UTSW.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven stage IV colon adenocarcinoma (any T [Tx, T1, T2, T3, or T4], N1- 2, M1). Tumors must be deemed to originate in the colon including tumors that extend into/involve the small bowel (e.g. those at the ileocecal valve).
2. Known DNA mismatch repair or microsatellite instability status. Only one of these tests is required for enrollment as there is 95% concordance rate of these tests.

   * The eligible patient's tumors be classified as proficient in DNA mismatch repair (pMMR) by immunohistochemistry (IHC) for MMR protein expression (MLH1, MutS homolog 2 (MSH2), MutS homolog 6 (MSH6), PMS2. Tumors with intact expression of all MMR proteins will be considered pMMR.
   * OR
   * The eligible patient's tumor be classified by Pathologic Complete Response (pCR) as stable microsatellite stability status (MSS) for panel of microsatellite markers, OR
   * MSS by commercially available next generation sequencing testing. OR
   * If tumor-based test are not feasible, then commercially available circulating tumor DNA tests showing MSS status will also be acceptable.
3. The patients should have received at least two lines of systemic chemotherapies in metastatic setting. They should have received fluoropyrimidine, irinotecan, and oxaliplatin unless medically contraindicated. Prior anti-VEGF (vascular endothelial growth factor) therapy is accepted for enrollment since anti-VEGF therapy maintains its benefit across several lines of therapy. If clinically appropriate, the patients should have received anti-EGFR (epidermal growth factor receptor) therapy for all Rat sarcoma (RAS) wild type colorectal cancers and v-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600E mutation-directed therapy for BRAF V600E mutant colorectal cancers and HER2 targeted therapy for HER2 amplified colorectal cancers.
4. Age 18 and above
5. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
6. Adequate organ and marrow function

   * Hemoglobin ≥ 9.0 g/dL
   * Lymphocyte count > 0.5 x 109/L (500/uL)
   * Absolute Neutrophil Count (ANC) ≥ 1500 mm3
   * Platelet Count ≥ 100,000 mm3
   * Creatinine ≤ 1.5 x upper limit of normal or Calculated Creatinine Clearance ≥ 45 mL/min
   * Total Bilirubin ≤ 1.5 x upper limit of normal unless Gilbert syndrome with the following exception: Patients with known Gilbert disease: serum bilirubin >3 ULN
   * Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) ≤ 2.5 x upper limit of normal
   * The subject's urinary protein is < 1+ on dipstick or routine urinalysis; if urine protein (which is equal to 30 mg/dL on random urine protein assessment); if urine protein is ≥ 2+ (equal to 100mg/dL on random urine protein assessment), a 24-hour urine must be collected and must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study.
   * Serum albumin ≥ 25 g/L (2.5 g/dL)
7. Negative HIV testing at screening, with following exception: patients with positive HIV tests at screening are eligible provided they are stable on anti-retroviral therapy, have a cluster of differentiation 4 (CD4) count > 200/uL, and have undetectable viral load.
8. Negative hepatitis B surface antigen (HBsAg) test at screening. If a prior testing is available within previous 12 months and negative, this criteria can be considered to be met.
9. Ability to understand and the willingness to sign a written informed consent
10. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control with <1% failure rate, tubal ligation, male sterilization; abstinence) prior to study entry, for the duration of study participation, and for 6 months following completion of therapy. Women must refrain from donating eggs during this same period. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months).
12. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening The HCV RNA test must be performed for patients who have a positive HCV antibody test. If a prior testing is available within previous 12 months and negative, this criteria can be considered to be met.

Exclusion Criteria:

1. Microsatellite unstable colorectal (MSI-H) cancers identified by PCR testing OR by commercially available Next-generation sequencing (NGS) and Circulating tumor DNA (ctDNA) testing OR by loss of expression of one or more of the MMR enzymes (MLH1, MSH2, MSH6, PMS2) on immunohistochemistry. Only one such test is required to confirm eligibility.
2. Current active known or suspected autoimmune disease such as including colitis, inflammatory bowel disease (i.e. ulcerative colitis or Crohn's disease), rheumatoid arthritis, pan-hypopituitarism, History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan, adrenal insufficiency treated with immunosuppressive steroids and biologics treatment. Patients with controlled disease with no active treatment or prednisone < 10 mg daily may be eligible based on treating physician assessment.

   Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, history of radiation pneumonitis in the radiation field (fibrosis) is permitted or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
3. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalent are permitted (although not encouraged) in the absence of active autoimmune disease.
4. Prior use of atezolizumab or ATRA is not eligible. Prior use of any other immunotherapy such anti programmed death-ligand 1 (PD-L1), anti- programmed cell death protein 1 (PD-1), Anti-CTLA4 will also be excluded.
5. Chemotherapy, radiotherapy, or other cancer therapy within 3 weeks prior to starting study treatment.
6. Subjects must have recovered from prior treatment-related to toxicities to grade 1 or baseline (excluding alopecia and clinically stable toxicities requiring ongoing medical management, such as hypothyroidism from prior immune checkpoint inhibitor treatment).
7. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study within 28 days prior to initiation of study treatment
8. Untreated brain metastases are not allowed. If prior treatment of brain metastases with surgery and/or radiation therapy has been provided, those patients will be clinically stable and not requiring escalating doses of steroids.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ATRA, atezolizumab, and bevacizumab or other agents used in study.
10. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), history of hypertensive crisis or hypertensive encephalopathy. Clinically significant cardiovascular disease, such as cerebrovascular accident within six months prior to enrollment, myocardial infarction within six months of prior to enrollment, unstable angina History of hypertensive crisis or hypertensive encephalopathy. If patient has previously received bevacizumab safely after that episode, with adequate BP control, then patients will be eligible.
11. Uncontrolled inter current illness including, but not limited to, ongoing or severe infection within 4 weeks prior to initiation of study treatment that could impact patient safety, symptomatic congestive heart failure with reduced ejection fraction history and the New York Heart Association (NYHA) Functional Classification class III or IV, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
12. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants. or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months for atezolizumab and 6 month for bevacizumab after the final dose of study treatment.

    Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
13. History of leptomeningeal disease or un-controlled tumor related pain. Patient requiring pain medications should be on a stable regimen. Symptomatic lesions (e.g. bone metastasis or metastasis causing nerve impingement) amenable to radiation therapy should be treated before enrollment and patient should have recovered from that radiation. No required minimum recovery period from the radiation.
14. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
15. Prior allogeneic stem cell or solid organ transplantation
16. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
17. History of Grade 4 venous thromboembolism. If previously have received bevacizumab safely after that episode then patients will be eligible
18. History of Grade > 2 hemoptysis (defined as > 2.5 mL of bright red blood per episode) within 1 month prior to screening
19. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
20. Currently active abdominal fistula, GI perforation, intra-abdominal abscess, or active GI bleeding requiring transfusion of blood products or hospitalization within 6 months
21. Serious, non-healing wound, active non-healing ulcer, or untreated bone fracture
22. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
23. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
24. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL or corrected serum calcium >ULN)
25. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
26. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
27. Known active hepatitis B or C, active tuberculosis and known uncontrolled HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of of ATRA, bevacizumab and atezolizumab combination | From time of enrollment/treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the objective response rate of ATRA, bevacizumab and atezolizumab combination. Complete response+ partial response measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in refractory microsatellite stable (proficient mismatch repair) colorectal cancers

SECONDARY OUTCOMES:
Disease Control Rate of of ATRA, bevacizumab and atezolizumab combination | From time of enrollment/treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the disease control rate of ATRA, bevacizumab and atezolizumab combination in microsatellite stable (proficient mismatch repair) colorectal cancers. Disease control rate (complete response+ partial response + stable disease) by using RECIST 1.1.
Frequency of adverse events | From time of enrollment/treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the safety of the combination treatment of ATRA, bevacizumab and atezolizumab combination in microsatellite stable (proficient mismatch repair) colorectal cancers by documenting the Frequency of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Kazmi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States